CLINICAL TRIAL: NCT07120204
Title: Evaluation of Radiofrequency Thermocoagulation Versus Corticosteroid Injection in Patients With Chronic Calcaneal Spur Related Plantar Fasciopathy Using Elastography and Foot Function Index
Brief Title: One Cause of Heel Pain is Plantar Fasciopathy (PF). In Most Cases, a Heel Spur is Frequently Present Alongside PF. We Aim to Evaluate the Efficacy of Corticosteroid Injection and Radiofrequency Ablation, Along With Tissue Elasticity Assessed by Ultrasound, in Patients With Chronic Pain (≥6 Months).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gülen Güler, Professor Doctor, Head of Anesthesiology and Reanimation Deparment, Head of Algology Department, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/60
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Plantar Fasciopathy; Chronic Pain; Corticosteroid Injection; Radiofrequency Ablation; Elasticity Imaging Techniques
Keywords: plantar fasciopathy; plantar fasciitis; randomized; radiofrequency thermal coagulation; RF; shear wave; elastography
MeSH Terms: conditions — Chronic Pain; Fasciitis, Plantar | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid Injection (Active Comparator): The patient will be in the lateral decubitus position with the symptomatic foot below. The symptomatic foot will be prepared with povidone-iodine and draped in a sterile manner. A sterile-covered ultrasound probe will be placed over the heel to visualize the calcaneus, plantar fascia, and any calcaneal spur. Subsequently, 1 mL of triamcinolone acetonide 40 mg (KENACORT-A IM/Intra-articular Retard 40 mg ampoule) and 1 mL of 2% lidocaine (Aritmal 2% ampoule) will be injected over the plantar fascia.
  Interventions: Drug: Corticosteroid Injection
- Radiofrequency Thermocoagulation (Active Comparator): The patient will be in the lateral decubitus position with the symptomatic foot below. The foot was prepared with povidone-iodine and draped under sterile conditions. A sterilized ultrasound probe was placed over the heel to visualize the calcaneus, plantar fascia, and calcaneal spur. A 10 cm long radiofrequency (RF) needle with a 5 mm active tip was advanced in-plane under ultrasound guidance toward the tip of the calcaneal spur. Sensory stimulation at 50 Hz elicited paresthesia in the medial calcaneus, while motor stimulation at 2 Hz did not produce any muscle contractions. The RF generator (Beijing Neo Science Co., RFE 4b) was set to 80 °C for 90 seconds, and the RFA procedure was initiated.
  Interventions: Procedure: Radiofrequency thermocoagulation

INTERVENTIONS:
Drug: Corticosteroid Injection — The symptomatic foot will be prepared with povidone-iodine and draped in a sterile manner. A sterile-covered ultrasound probe will be placed over the heel to visualize the calcaneus, plantar fascia, and any calcaneal spur. Subsequently, 1 mL of triamcinolone acetonide 40 mg (KENACORT-A IM/Intra-articular Retard 40 mg ampoule) and 1 mL of 2% lidocaine (Aritmal 2% ampoule) will be injected over the plantar fascia.
  Arms: Corticosteroid Injection
Procedure: Radiofrequency thermocoagulation — The patient will be in the lateral decubitus position with the symptomatic foot below. The foot was prepared with povidone-iodine and draped under sterile conditions. A sterilized ultrasound probe was placed over the heel to visualize the calcaneus, plantar fascia, and calcaneal spur. A 10 cm long radiofrequency (RF) needle with a 5 mm active tip was advanced in-plane under ultrasound guidance toward the tip of the calcaneal spur. Sensory stimulation at 50 Hz elicited paresthesia in the medial calcaneus, while motor stimulation at 2 Hz did not produce any muscle contractions. The RF generator (Beijing Neo Science Co., RFE 4b) was set to 80 °C for 90 seconds, and the RFA procedure was initiated.
  Arms: Radiofrequency Thermocoagulation

SUMMARY:
Heel pain is common among adults. One cause of heel pain is plantar fasciopathy (PF). In most cases, a heel spur, a bony prominence that extends into the plantar fascia, is frequently present alongside PF. First-line treatments include pain-relieving drugs, home exercises, heel support peds, and physical therapy. However, some patients can't get relief from these therapies, and the pain persists beyond six months. This situation is referred to as refractory chronic PF. Local treatments applied via skin puncture such as anti-inflamtory injection and destruction of nerves carrying pain signals to brain are warranted in these cases. We aim to evaluate the efficacy of corticosteroid injection and radiofrequency ablation, along with tissue elasticity assessed by ultrasound, in patients with chronic pain (≥6 months).

The goal of this clinical trial is to determine which treatment-corticosteroid injection or radiofrequency thermal thermocoagulation-is more effective for treating plantar fasciopathy in adults. It will also learn about the effects of the treatments on the properties of the heel tissue using ultrasound. The main questions it aims to answer are:

Do corticosteroid injections and radiofrequency thermal thermocoagulation have the same efficacy on pain and functionality for both short- and long-term? Do corticosteroid injections and radiofrequency thermal thermocoagulation similarly affect heel tissue? The researchers will investigate which of the corticosteroid injection and radiofrequency thermocoagulation is more effective for

DETAILED DESCRIPTION:
Plantar fasciopathy (PF) is one of the most common causes of foot pain, accounting for approximately 10-15% of all cases. The plantar fascia originates from the calcaneus on the plantar surface of the foot and inserts into the proximal phalanges. It becomes tense while standing and provides support to the medial longitudinal arch. Although the pathophysiology of PF is not fully understood, repetitive mechanical overload is believed to cause microtears, particularly at the medial origin of the plantar fascia. Subsequent inflammation and degeneration may become chronic, and excessive traction at the medial calcaneus can lead to the formation of a bony outgrowth called a calcaneal spur. This bony protrusion may increase pain by causing inflammation, nerve compression, and atrophy of the heel fat pad. Approximately 67% of patients with PF present with a calcaneal spur.

Typically, patients complain of heel pain upon taking their first steps in the morning or after periods of rest, and during weight-bearing activities. On physical examination, tenderness is usually observed along the medial aspect of the heel, and pain is exacerbated with toe extension. Diagnosis is generally based on clinical history and physical examination. Ultrasound imaging can aid in diagnosis due to its rapid application and bedside availability. Conventional ultrasonography may reveal thickening of the plantar fascia, perifascial edema, hypoechoic areas within the fascia, and the presence of a calcaneal spur.

Shear wave elastography (SWE) is a modern, non-invasive ultrasound modality that measures tissue stiffness and elasticity. Measuring the stiffness of the plantar fascia using SWE, along with B-mode parameters, can facilitate diagnosis. Moreover, it allows monitoring of structural changes in the fascia following treatment.

Treatment options for PF include non-steroidal anti-inflammatory drugs (NSAIDs), physical therapy, orthotics, night splints, corticosteroid injections (CSIs), platelet-rich plasma injections, extracorporeal shockwave therapy, and radiofrequency ablation (RFA). While corticosteroid injection may provide short-term pain relief, it is associated with risks, including alteration of connective tissue microstructure and fat pad atrophy. In RFA, continuous electrical current generates heat, leading to the destruction of nociceptive free nerve endings in the target area. RFA has been successfully used for decades in the management of lower back pain, head and facial pain, sympathetic chain ablation, and joint pain. Various studies have also supported its efficacy and safety in treating PF.

The primary aim of this study is to compare the effectiveness of RFA and CSI using the Foot Function Index (FFI) score at 6 months. The secondary aim is to assess pain scores and structural changes in the plantar fascia using SWE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic (≥ 6 months) plantar fasciopathy
2. NRS score ≥ 4
3. Presence of a calcaneal spur detected by ultrasound (USG) or direct radiography
4. At least one of the following treatments has been administered:

   * Home exercise program
   * Physiotherapy
   * Orthosis/prosthesis
   * NSAIDs
   * Night splint
   * Kinesio taping
   * Corticosteroid injection
   * Extracorporeal shock wave therapy (ESWT)

Exclusion Criteria:

1. History of calcaneal trauma/fracture
2. Previous radiofrequency ablation (RFA) treatment
3. Patients with seronegative spondyloarthropathy
4. Inflammatory or degenerative arthropathies
5. Presence of diabetes
6. Pregnancy
7. History of cancer
8. Peripheral neuropathy or ischemia
9. Open wound or signs of infection at the procedure site
10. Evidence of systemic infection
11. Patients using anticoagulant or antiplatelet agents
12. Presence of an intracardiac defibrillator or pacemaker
13. Patients with tarsal tunnel syndrome
14. Patients who have received ESWT and/or corticosteroid injection within the last 3 months
15. Presence of heel pain due to lumbar radiculopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Foot Function Index Score (FFI) | 6 months after treatment
  FFI includes 23 11-point Likert-type questions about feet. The lowest score is 0, and the highest score is 100. A lower score is better.

SECONDARY OUTCOMES:
Numeric Rating Scale-11 (NRS-11) Scores | 6 months after treatment
  NRS-11 is an 11-point Likert-type scale that assesses pain severity. The lowest score is 0, and the highest score is 10. A lower score is better

OTHER OUTCOMES:
Foot Function Index (FFI) | 1 month after treatment
  FFI includes 23 11-point Likert-type questions about feet. The lowest score is 0, and the highest score is 100. A lower score is better
Foot Function Index (FFI) | Baseline
  FFI includes 23 11-point Likert-type questions about feet. The lowest score is 0, and the highest score is 100. A lower score is better
Foot Function Index (FFI) | 3 months after treatment
  FFI includes 23 11-point Likert-type questions about feet. The lowest score is 0, and the highest score is 100. A lower score is better
Numeric Rating Scale-11 (NRS-11) Scores | Baseline
  NRS-11 is an 11-point Likert-type scale that assesses pain severity. The lowest score is 0, and the highest score is 10. A lower score is better
Numeric Rating Scale-11 (NRS-11) Scores | 1 month after treatment
  NRS-11 is an 11-point Likert-type scale that assesses pain severity. The lowest score is 0, and the highest score is 10. A lower score is better
Numeric Rating Scale-11 (NRS-11) Scores | 3 months after treatment
  NRS-11 is an 11-point Likert-type scale that assesses pain severity. The lowest score is 0, and the highest score is 10. A lower score is better

CONTACTS AND LOCATIONS:
Overall Officials: Gülen Güler, Prof. Dr., M.D., Study Director — Erciyes Üniversity School of Medicine, Anesthesiology and Reanimation Department
Locations (1):
- Erciyes Üniversitesi Tıp Fakültesi, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Deindividualized data will be shared upon reasonable request.
Supporting Information: SAP, ICF
Time Frame: 1 year after the study is completed.

REFERENCES:
- [Background] Neufeld SK, Cerrato R. Plantar fasciitis: evaluation and treatment. J Am Acad Orthop Surg. 2008 Jun;16(6):338-46. doi: 10.5435/00124635-200806000-00006. PMID 18524985